CLINICAL TRIAL: NCT00704899
Title: Effect of Anti-Depressants vs Physiotherapy in Management of Fibromyalgia Syndrome: What Predicts a Clinical Benefit?
Brief Title: Anti-Depressants vs Physiotherapy in Management of Fibromyalgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mahatma Gandhi Institute of Medical Sciences (Other)
Responsible Party: Prof AP Jain, Department of Medicine, MGIMS Sevagram
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MGIMS-001
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Last update posted 2008-07-04 (Estimated); Status verified 2008-06

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Experimental): anti-depressants
  Interventions: Drug: Amitryptiline
- 1 (Experimental): physiotherapy
  Interventions: Procedure: Physiotherapy

INTERVENTIONS:
Procedure: Physiotherapy — Structured exercise regimen
  Arms: 1
Drug: Amitryptiline — Amitryptiline 25mg once daily
  Arms: 2

SUMMARY:
To compare the efficacy of physiotherapy and anti-depressants in disability reduction in patients of Fibromyalgia syndrome.

DETAILED DESCRIPTION:
Research Question:

Does the use of physiotherapy or pharmacotherapy help in improving quality of life in patients of fibromyalgia as judged by fibromyalgia impact questionnaire at a 6 month follow up period?

Study hypothesis:

Physiotherapy is no better than pharmacotherapy in improving the quality of life in patients of fibromyalgia as judged by fibromyalgia impact questionnaire.

Study type- Interventional STUDY DESIGN: open label alternate patient treatment allocation Ethical approval for the trial protocol has been obtained from the institute's ethics committee of Mahatma Gandhi Institute of Medical Sciences, Sevagram.

Subjects and Methods The study will be conducted in Kasturba Hospital and Mahatma Gandhi Institute of Medical Sciences, Sevagram, from 1 march 2006 - 1 dec 2007. Patients will be selected to enter the study, in such a way that every patient presenting with chronic muscular pain will be screened in the study and patients fulfilling inclusion criteria will be recruited in the study.

Study population:

Total of 175 patients will be included in the study.

Methods:

The investigators will screen all patients who are referred to them for inclusion in the study. Written informed consent will be obtained from all participants. The patients included in the study will be administered a standardized questionnaire to record socio-demographic characteristics, symptom characteristics and history of previous visits to a health care provider. The socio-economic score (SES) will be determined using a validated questionnaire.[6] Briefly, the questionnaire consists of following: (1) household profile, (2) material possession profile, (3) educational profile, (4) occupational profile, (5) economic profile (6) possessed land or house cost profile and (7) social profile. Fibromyalgia impact questionnaire (FIQ) will be used to determine a baseline score. [7] For the purpose of the study this questionnaire is translated to local language (Marathi), and back-translated to English to ensure its accuracy. Minor modifications have been done in the questionnaire to make it suitable for our setting (for example: the use of washer or dryer for laundry was modified to washing the laundry by themselves). Assessment of psychiatric co morbidity will be done using the Brief Psychiatric Rating Scale (BPRS), which is an 18 item instrument, each item has a seven severity grades.[8] A score of 32 or more indicates presence of psychopathology.[9]

Interventions:

A trained Physiotherapist will conduct a uniform structured physical training and aerobic session for one group of patients. The patients will be advised to perform the exercises daily twice for at least 10 minutes. There will be a step up pattern of exercise regimen followed with relaxation, stretching and strengthening techniques. The methodology is described in box 1. The second group of patients will receive antidepressant in the form open label amitriptyline 25 mg once daily at bedtime. The dose of the drug may be increased if required. All patients will be also offered pharmacologic treatment with 50 mg tramadol in thrice daily doses and as required. The treatment recommendations are based on standard recommendations on the management of fibromyalgia.[5]

Outcome assessment All patients will be followed up for six months at monthly intervals. At each visit the study investigators will determine the course of the disease and compliance with therapy. The FIQ score will be assessed at the end of 6 monthly visits. Reduction in FIQ score from the baseline will be used as the principle outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Patient's between 18-60 yrs, belonging to either sex. With symptoms of chronic muscular pain of at least 12 weeks (that may or may not be consecutive) who fulfill the American College of Rheumatology (ACR) criteria for the diagnosis of Fibromyalgia

Exclusion Criteria:

* Patients of age group more than 60 yrs and below 18 years
* Pregnant or lactating females.
* Patients with a history of trauma.
* Patients with severe co morbid illness which prevents physical activity (for example, cardiovascular problems)
* Patients with the presence of specific medical disorders which require immediate treatment (for example, fractures, infectious diseases),
* Patients with associated neurological abnormality

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 175 (Actual)
Dates: Start 2006-03; Primary Completion 2007-12 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Reduction in FIQ score from the baseline | Two years

SECONDARY OUTCOMES:
Reduction in Tender point score | Two years
Reduction in Brief psychiatric rating score | Two Years

CONTACTS AND LOCATIONS:
Locations (1):
- Mahatma Gandhi Institute of Medical Sciences, Sevāgrām, Maharashtra, India